CLINICAL TRIAL: NCT05439031
Title: StereoTactic Arrhythmia Radiotherapy in the NetherLands no. 2
Acronym: STARNL-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Heart Foundation (Other)
Responsible Party: Principal Investigator, Pieter G. Postema, Principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL80617.018.22
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Ventricular Tachycardia; Arrythmia, Cardiac
Keywords: Ventricular Arrhythmias; Ventricular Tachycardia; Cardiac Radioablation; Stereotactic Radiotherapy; Stereotactic Arrhythmia Radiotherapy; Stereotactic body radiotherapy; Cardiac ablative radiotherapy
MeSH Terms: conditions — Tachycardia, Ventricular; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Arrhythmia Radiotherapy (Experimental): Patients will undergo stereotactic arrhythmia radiotherapy and subsequent follow-up.
  Interventions: Radiation: Stereotactic Arrhythmia Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Arrhythmia Radiotherapy — Single radiation treatment of 25 Gy with external beam radiation therapy to the pro-arrhythmic region as determined by the cardiologist-electrophysiologist and radiation-oncologist combined
  Other Names: Cardiac Radioablation

SUMMARY:
Ventricular tachycardia (VT) is a malignant cardiac arrhythmia subjecting our patients to a high risk of sudden death, increased morbidity and reduced quality of life. Unfortunately, failure of treatment is common and VT recurrences remain an important concern. In these patients, stereotactic arrhythmia radiotherapy appears to be an effective and safe treatment. The mechanism of action however remains unknown and should be elucidated.

The objective of this phase 2, single arm, monocenter, pre-post intervention study is to evaluate the efficacy and safety of stereotactic arrhythmia radiotherapy and obtain insights in the mechanism of action by evaluating electro-anatomical alterations of stereotactic arrhythmia radiotherapy in patients with therapy refractory ventricular tachycardia.

DETAILED DESCRIPTION:
Ventricular tachycardia (VT) is a malignant cardiac arrhythmia leading to a sudden abolition of cardiac function directly followed by a shortage of oxygen supply to essential organs such as the brain and heart. For this reason, VT is a cardiac emergency and should be treated within seconds to minutes before irreversible and potentially fatal organ damage follows. Current treatment options are limited to anti-arrhythmic drugs, an implantable cardioverter defibrillator (ICD), and invasive catheter ablation. Unfortunately, invasive cardiac VT ablation has the lowest success rate and the highest complication rates among all arrhythmia ablations.

Since the first case series published by Cuculich et al. (2017) and the first prospective trial published by Robinson et al. (2019), stereotactic arrhythmia radiotherapy (STAR) has evolved as a new treatment modality for patients with ventricular tachycardia refractory to conventional therapies. Patients are treated with a single radiotherapy fraction of 25 Gy at the determined pro-arrhythmic cardiac region with the use of standard stereotactic radiotherapy techniques. Experience with STAR is steadily growing worldwide. In the systematic review by Van der Ree et al. (2020), a reduction of >85% in VT episodes with a simultaneously promising safety profile was shown.

The mechanism of action of STAR is not yet fully known and is yet to be elucidated. The pathophysiological mechanism of VT relies on re-entry due to zigzag conduction by the surviving myocardial fibers in previously damaged heart tissue. At first, it was hypothesized that inducing cell-death by ionizing radiation leads to dense transmural fibrosis. As mature myocardial fibrosis is not able to propagate electrical activation this may lead to the abolishment of the zigzag conduction herewith reducing the chance of re-entry and VT. Fibrosis maturation takes several weeks to months to complete. However, the anti-arrhythmic effects seem to occur earlier. In preclinical studies, early electrophysiological alterations were demonstrated (Zhang et al. 2021). The gap-junction protein connexion-43 (Cx43) and the voltage gated sodium channels were upregulated, leading to a supraphysiological state with increased conduction velocity. Since a slow conduction pathway is required for re-entry, this could explain the timing of the observed effect, although the exact mechanism of action remains to be elucidated.

In the STARNL-2 study we aim to confirm our STARNL-1 pilot (6 patients) efficacy and safety data in a larger cohort and obtain insights in the electro-anatomical alterations of stereotactic arrhythmia radiotherapy in patients with therapy refractory ventricular tachycardia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Implanted ICD
* World Health Organization (WHO) / Eastern Cooperative Oncology Group (ECOG) performance status grade 0-3 in the past 3 months (from fully active to capable of limited self-care, see below for full explanation)
* At least 3 episodes of treated VT within the last 3 months
* Recurrence of VT after

  * Failed or intolerant to least one class 1 or class 3 anti-arrhythmic drug AND
  * At least one catheter ablation procedure OR considered to be unsuitable for a catheter ablation procedure (e.g. no sufficient vascular access, considered unfit to undergo prolonged general anesthesia, comorbid conditions resulting in unacceptable peri-procedural risks)
* Able and willing to undergo all necessary evaluations, treatment and follow-up for the study and of follow-up thereafter

Exclusion Criteria:

* Pregnancy
* History of radiation treatment in the thorax or upper abdominal region
* Interstitial pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in the number of treated VT episodes | 18 months (excluding 3 months of blanking period)
  The main efficacy measure is a reduction in the number of treated VT episodes by ≥50% at the end of follow-up of 1 year (including a blanking period of 3 months). Net follow-up is 9 months compared to 9 months before treatment.
Rate of treatment related serious adverse events (SAEs) | 12 months
  The main safety measure is defined by a ≤20% rate of treatment related serious adverse events (SAEs), determined as the number of treatment related serious adverse events per number of treatment related adverse events.

SECONDARY OUTCOMES:
Reduction in the number of treated and non-treated VT episodes | 18 months (excluding 3 months of blanking period)
  Reduction in the number of treated and non-treated VT episodes by ≥70% at the end of follow-up compared to the year before treatment.
Reduction in anti-arrhythmic drugs | 12 months
  A reduction of the daily dose by ≥50% (amiodarone or mexiletine) at the end of follow-up compared to baseline.
Quality of Life improvement | 12 months
  Quality of life improvement of ≥25% in the categories health change and social functioning as measured by the SF-36 questionnaire at the end of follow-up compared to baseline.
Cardiac safety | 12 months
  >25% relative decrease in left ventricular ejection fraction measured by echocardiography at end of follow-up as compared to baseline
Pulmonary safety | 12 months
  >25% relative decrease in forced expiratory volume in 1 second (FEV1) measured by pulmonary functions tests at end of follow-up as compared to baseline.
Pulmonary safety | 12 months
  >25% relative decrease in diffusing capacity (DLCO) measured by pulmonary functions tests at one year after treatment as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pieter G Postema, MD PhD, Principal Investigator — University of Amsterdam
Locations (1):
- Amsterdam UMC location University of Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cuculich PS, Schill MR, Kashani R, Mutic S, Lang A, Cooper D, Faddis M, Gleva M, Noheria A, Smith TW, Hallahan D, Rudy Y, Robinson CG. Noninvasive Cardiac Radiation for Ablation of Ventricular Tachycardia. N Engl J Med. 2017 Dec 14;377(24):2325-2336. doi: 10.1056/NEJMoa1613773. PMID 29236642
- [Background] Robinson CG, Samson PP, Moore KMS, Hugo GD, Knutson N, Mutic S, Goddu SM, Lang A, Cooper DH, Faddis M, Noheria A, Smith TW, Woodard PK, Gropler RJ, Hallahan DE, Rudy Y, Cuculich PS. Phase I/II Trial of Electrophysiology-Guided Noninvasive Cardiac Radioablation for Ventricular Tachycardia. Circulation. 2019 Jan 15;139(3):313-321. doi: 10.1161/CIRCULATIONAHA.118.038261. PMID 30586734
- [Background] van der Ree MH, Blanck O, Limpens J, Lee CH, Balgobind BV, Dieleman EMT, Wilde AAM, Zei PC, de Groot JR, Slotman BJ, Cuculich PS, Robinson CG, Postema PG. Cardiac radioablation-A systematic review. Heart Rhythm. 2020 Aug;17(8):1381-1392. doi: 10.1016/j.hrthm.2020.03.013. Epub 2020 Mar 20. PMID 32205299
- [Background] Zhang DM, Navara R, Yin T, Szymanski J, Goldsztejn U, Kenkel C, Lang A, Mpoy C, Lipovsky CE, Qiao Y, Hicks S, Li G, Moore KMS, Bergom C, Rogers BE, Robinson CG, Cuculich PS, Schwarz JK, Rentschler SL. Cardiac radiotherapy induces electrical conduction reprogramming in the absence of transmural fibrosis. Nat Commun. 2021 Sep 24;12(1):5558. doi: 10.1038/s41467-021-25730-0. PMID 34561429